CLINICAL TRIAL: NCT00988208
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Docetaxel and Prednisone With or Without Lenalidomide in Subjects With Castrate-Resistant Prostate Cancer (CRPC)
Brief Title: Study to Evaluate Safety and Effectiveness of Lenalidomide in Combination With Docetaxel and Prednisone for Patients With Castrate-Resistant Prostate Cancer
Acronym: Mainsail
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-5013-PC-002; EudraCT Number 2008-007969-23
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Results first posted 2013-09-05 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Prostate Cancer
Keywords: Castrate-Resistant Prostate Cancer; Revlimid; Lenalidomide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lenalidomide; Docetaxel; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel, Prednisone, Lenalidomide (DPL) (Experimental): 25 mg lenalidomide orally once each day on Days 1-14; 75 mg/m2 docetaxel intravenously on Day 1; 5 mg prednisone orally twice daily on each day of the treatment cycle
  Interventions: Drug: Lenalidomide; Drug: Docetaxel; Drug: Prednisone
- Docetaxel and Prednisone (DP) (Experimental): Oral placebo once each day on Days 1-14 of the treatment cycle; 75 mg/m2 docetaxel intravenously on Day 1; 5 mg prednisone orally twice each day on each day of the treatment cycle
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: Placebo

INTERVENTIONS:
Drug: Lenalidomide — 25 mg lenalidomide orally once each day on Days 1-14
  Other Names: CC-5013; Revlimid
  Arms: Docetaxel, Prednisone, Lenalidomide (DPL)
Drug: Docetaxel — 75 mg/m2 intravenous docetaxel on Day 1
  Other Names: Taxotere
Drug: Prednisone — 5 mg prednisone orally twice daily on each day of the treatment cycle
  Other Names: There are multiple brand names for prednisone.
Drug: Placebo — Oral placebo once each day on Days 1-14 of the treatment cycle
  Arms: Docetaxel and Prednisone (DP)

SUMMARY:
The purpose of the study is to determine whether lenalidomide is safe and effective for use in combination with docetaxel and prednisone for the treatment of subjects with metastatic Castrate-Resistant Prostate Cancer.

The addition of lenalidomide to docetaxel and prednisone is proposed to increase the life expectancy of these subjects.

DETAILED DESCRIPTION:
In November 2011, the Data Monitoring Committee concluded it was unlikely that the study would meet its primary endpoint of overall survival (OS) and recommended that the study be stopped. The study was terminated in accordance with this recommendation. All sites were instructed to immediately discontinue all patients from experimental lenalidomide/placebo treatment administered either in combination with chemotherapy or as a single agent following chemotherapy discontinuation. Subsequently, Protocol Amendment 3 was issued to provide for the following:

To continue to collect information on Second Primary Malignancies (SPMs) and additional treatments for Prostate Cancer in all randomized subjects during survival follow-up.

To continue to provide docetaxel and prednisone for up to 10 cycles to subjects randomized at non-US sites who were ongoing in the CC-5013-PC-002 protocol when the decision was made to discontinue lenalidomide/placebo and who were experiencing benefit as per investigator discretion. For subjects who had exceeded 10 cycles of docetaxel and prednisone at the time of Protocol Amendment 3 approval, an additional two cycles were provided.

All references to dosing and study procedures pertaining to the safety, efficacy, and exploratory endpoints of lenalidomide/placebo were discontinued as part of Protocol Amendment 3.

ELIGIBILITY:
Inclusion Criteria:

1. Must sign an Informed Consent Form (ICF)
2. Males ≥ 18 years of age
3. Able to adhere to the study visit schedule and requirements of the protocol
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
5. Life expectancy of ≥ 12 weeks
6. Willingness to participate in Patient-Reported Outcomes assessments
7. Serum testosterone levels < 50 ng/dL
8. Confirmed metastatic adenocarcinoma of the prostate that is unresponsive or refractory to hormonal therapy
9. Have documented disease progression while receiving or following hormonal therapy as determined by increasing Serum Prostate Specific Antigen (PSA) level, Radiological Progression, or ≥2 new bone lesions
10. Subjects must agree to receive counseling related to pregnancy precautions, teratogenic and other risks of lenalidomide
11. Refrain from donating blood or semen as defined by protocol

Exclusion Criteria:

1. A history of clinically significant disease that places subject at an unacceptable risk for study entry
2. Prior Therapy with thalidomide, lenalidomide or pomalidomide
3. Prior chemotherapy for prostate cancer
4. Use of any other experimental drug or therapy within 28 days prior to randomization
5. Prior radiation to ≥ 30% of bone marrow or any radiation therapy within 28 days prior to randomization
6. Prior use of Strontium-89 at any time or Samarium-153 within 56 days prior to randomization
7. Surgery within 28 days prior to randomization
8. Concurrent anti-androgen therapy
9. Abnormal serum chemistry or hematology laboratory values
10. Significant active cardiac disease within the previous 6 months:
11. Thrombotic or thromboembolic events within the past 6 months:
12. History of peripheral neuropathy of ≥grade 2
13. History of severe hypersensitivity reaction to drugs formulated with polysorbate 80
14. Paraplegia
15. History of Central nervous system (CNS) or brain metastases
16. History of malignancies other than prostate cancer within the past 5 years, with the exception of treated basal cell/squamous cell carcinoma of the skin
17. Concurrent use of alternative cancer therapies

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1059 (Actual)
Dates: Start 2009-11-11 (Actual); Primary Completion 2012-01-13 (Actual); Study Completion 2016-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debora Barton, MD, Study Director — Celgene Corporation
Locations (210):
- United States (66):
  - Hematology Oncology Associates, Phoenix, Arizona
  - Northern AZ Hematology and Oncology Assoc, Sedona, Arizona
  - Arizona Oncology, Tucson, Arizona
  - City of Hope Cancer Center, Duarte, California
  - Southwest Cancer Center - Escondido, Escondido, California
  - Scripps Cancer Center - Clinical Research, La Jolla, California
  - VA Long Beach Healthcare System, Long Beach, California
  - The Angeles Clinc and Research Institute, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Prostate Oncology Specialists, Marina del Rey, California
  - Stanford University Medical Center, Stanford, California
  - Rocky Mountain Cancer Centers-Colorado Springs Circle, Colorado Springs, Colorado
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - Advanced Medical Specialties, Miami, Florida
  - Florida Cancer Institute - New Hope, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida, P.A.- West Gore Street, Orlando, Florida
  - South Florida Oncology - Hematology, Tamarac, Florida
  - Palm Beach Cancer Institute, LLC, West Palm Beach, Florida
  - Cancer Care and Hematology Specialists of Chicagoland, Niles, Illinois
  - Lutheran General Hospital, Park Ridge, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - Hematology and Oncology Specialist, LLC, Metairie, Louisiana
  - Maryland Oncology Hematology PA, Columbia, Maryland
  - Minnesota Oncology Hematology, PA, Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Summit Medical Group Overlook Oncology Center, Berkeley Heights, New Jersey
  - Hematology-Oncology Associates of NNJ, P, Morristown, New Jersey
  - Hematology Oncology Associates of South Jersey, Mount Holly, New Jersey
  - New York Oncology Hematology P.C., Albany, New York
  - Columbia Univ Medical Center, New York, New York
  - Weill Cornell Medical College Dr. Feldman's Office, New York, New York
  - New Bern Cancer Care, New Bern, North Carolina
  - Cancer Centers of North Carolina, Raleigh, North Carolina
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Northwest Cancer Specialists-Tualatin, Tualatin, Oregon
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Cancer Center of the Carolinas, Greer, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Sarah Cannon Research Institute UK, Nashville, Tennessee
  - Texas Oncology, P.A.-Amarillo, Amarillo, Texas
  - Texas Oncology-Arlington South, Arlington, Texas
  - Texas Oncology, PA, Austin, Texas
  - Baylor Sammons Cancer Center, Dallas, Texas
  - Texas Oncology, P.A.-Fort Worth, Fort Worth, Texas
  - Longview Cancer Center, Longview, Texas
  - Allison Cancer Center, Midland, Texas
  - Texas Oncology, P.A. - Paris, Paris, Texas
  - Southlake Oncology, Southlake, Texas
  - Texas Oncology, P.A. - Tyler, Tyler, Texas
  - Texas Oncology Deke Slayton Cancer Center, Webster, Texas
  - Texas Oncology-Texoma Cancer Center, Wichita Falls, Texas
  - Veterans Education and Research Association of Northern New England, Inc., White River Junction, Vermont
  - Cancer Outreach Associates, Abingdon, Virginia
  - Fairfax Northern Virginia Hematology Oncology, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - Columbia Basin Hematology and Oncology, Kennewick, Washington
  - VA Puget Sound HCS Seattle Division, Seattle, Washington
  - Evergreen Hematology and Oncology, Spokane, Washington
- Australia (13):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
  - Flinders Medical Centre, Bedford Park
  - Chris O'Brien Lifehouse, Camperdown
  - Sir Charles Gairdner Hospital, Nedlands
  - Port Macquarie Base Hospital, Port Macquarie
  - Redcliffe Hospital, Redcliffe
  - Royal North Shore Hospital, St Leonards
  - Newcastle Calvary Mater Hospital, Waratah
  - Westmead Hospital, Westmead
  - Border Medical Oncology, Wodonga
  - The Queen Elizabeth Hospital, Woodville South
  - Princess Alexandra Hospital, Woolloongabba
- Austria (4):
  - Medical University of Graz, Graz
  - Landeskrankenhaus Salzburg, Salzburg
  - Krankenhaus der Barmherzigen Brueder, Vienna
  - Medizinische Universitat Wien, Vienna
- Belgium (6):
  - ZNA Middelheim, Antwerp
  - Hopital Erasme, Brussels
  - Edith Cavell Clinic, Brussels
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - AZ Nikolaas, Sint-Niklaas
- Canada (2):
  - The Health Institute for Men CMX Research Inc, Toronto, Ontario
  - Les Urologues Specialises, Montreal, Quebec
- Czechia (3):
  - Krajska zdravotni, a.s. Nemocnice Chomutov, o.z., Chomutov
  - Fakultni nemocnice Motol, Prague
  - Krajska zdravotni, a.s. - Masarykova nemocnice v Usti nad La, Ústí nad Labem
- Denmark (4):
  - Arhus Universitets hospital, Aarhus C
  - Rigshospitalet University Hospital, Copenhagen
  - Herlev Hospital, Herlev
  - Odense Universitetshospital, Odense C
- France (14):
  - CRLCC Paul Papin, Angers
  - Institut Bergonie Centre Regional de Lutte Contre Le Cancer de Bordeaux Et Sud Ouest, Bordeaux
  - Centre Georges Francois Leclerc, Dijon
  - Clinique Victor Hugo, Le Mans
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Clinique de Valdegour, Nîmes
  - CHU de Poitiers, Poitiers
  - Centre Eugene Marquis, Rennes
  - Institut de Cancerologie de la Loire, Saint Priest En Jaroz
  - CRLCC Centre Rene Gauducheau, Saint-Herblain
  - Hopital Civil de Strasbourg, Strasbourg
  - CHRU Hopital Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif
- Germany (14):
  - Vivantes Klinikum am Urban, Berlin
  - Medizinisches Zentrum Bonn-Friedensplatz, Bonn
  - Diakonissenkrankenhaus Dessau gGmbH, Dessau
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Krankenhaus Nordwest, Frankfurt a.M.
  - Onkologische Praxis Freiburg, Freiburg im Breisgau
  - Universitatsklinikum Hamburg-Eppendorf / IVDP, Hamburg
  - IORC- Innovation Onkologie Research and Consulting GmbH, Hamburg
  - Praxis fuer Haematologie und Onkologie Koblenz, Koblenz
  - Vituro GmbH & Co KG, Leipzig
  - TU München - Klinikum rechts der Isar, München
  - Universitaetsklinikum Muenster, Münster
  - University-Hospital Tübingen, Tübingen
  - Universitatsklinikum Ulm, Ulm
- Greece (4):
  - Alexandra General Hospital of Athens, Athens
  - Agioi Anargyroi Hospital, Athens
  - University Hospital of Larissa, Larissa
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Hungary (4):
  - Fovarosi Onkirmanyzat Peterfy S.Utcai Korhaz-Rend.Int es Baleseti Kozp., Budapest
  - Fovarosi Onkormanyzat Bajcsy-Zsilinszky Korhaz es Rendelointezet, Budapest
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Pecsi Tudomanyegytem Altalanos Orvostudomanyi Kar, Pécs
- Israel (4):
  - The Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center, Petah Tikva
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (10):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - Ordine Mauriziano, Candiolo
  - Azienda Ospedaliera Istituti Ospitalieri di Cremona, Cremona
  - Ospedale Vito Fazzi, Lecce
  - Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori (I.R.S.T.), Meldola
  - Ospedale di Mirano, Mirano (VE)
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedale degli Infermi di Rimini, Rimini
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Azienda Ospedaliero-Universitaria Santa Maria della Miserico, Udine
- Mexico (4):
  - Hospital Angeles Lindavista, D.F, DF
  - Consultorio de Especialidad en Urologia Privado, Durango, DGO
  - Hospital Fatima, Sinaloa, SIN
  - Consultorio Privado- Dr Jose Arturo Rodriguez Rivera, Zapopan, JAL
- Netherlands (16):
  - VU University Medical Center VU Medisch Centrum, Amsterdam
  - Ziekenhuis Rijnstate, Arhem
  - Amphia Ziekenhuis Molengracht, Breda
  - Gemini Ziekenhuis, Den Helder
  - Albert Schweitzer Ziekenhuis Amstelwijck, Dordrecht
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leids Universitair Medisch Centrum, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Erasmus Medical Center, Rotterdam
  - Erasmus Medisch Centrum, Rotterdam
  - HagaZiekenhuis, The Hague
  - Twee Steden Ziekenhuis Tilburg, Tilburg
  - VieCuri Medisch Centrum Venlo, Venlo
  - Isala Klinieken, Zwolle
- Poland (7):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Regionalny Osrodek Onkologiczny WSS im. M. Kopernika, Lodz
  - ZOZ MSWiA z Warminsko- Mazurskim Centrum Onkologii, Olsztyn
  - NZOZ Olsztynski Osr. Onkologiczny Kopernik Sp.z o.o, Olsztyn
  - SPZOZ Wojewodzki Szpital Specjalistyczny nr 3 w Rybniku, Rybnik
  - Centrum Onkologii-Instytut im.Marii Sklodowskiej-Curie, Warsaw
  - 4 Wojskowy Szpital Kliniczny z Poliklinika SP ZOZ, Wroclaw
- Russia (7):
  - Moscow Oncology Clinical Dispensary 1, Moscow
  - Medical Radiology Research Centre RAMS, Obninsk
  - State Institution of Heath Omsk Regional Oncology Dispensary, Omsk
  - Russian Scientific Center for Radiology and Surgical Technol, St. Petersburg, Pesochny Vlg Saint Petersburg
  - NSHI Dorozhnaya Clinical Hospital of OAO Russian Railways, Rostov-on-Don
  - Oncology Dispensary 2 of Krasnodar Region, Sochi
  - Yaroslavl Regional Clinical Oncology Hospital, Yaroslavl
- South Africa (6):
  - Groote Schuur Hospital, Cape Town, W Cape
  - The Oncology Centre Durban, Durban, KZ-Natal
  - Westridge Medical Centre, Durban, KZ-Natal
  - Netcare Oncology and Interventional Centre, Goodwood, W Cape
  - Dr. H. Malan, Polokwane
  - Pretoria Urology Hospital, Pretoria
- Spain (9):
  - Hospital del Mar, Barcelona
  - Hospital Durán i Reynals - Instituto Catalàn de Oncologìa ICO, Hospitalet de Llobregat, Barcelona
  - Hospital Arnau de Vilanova, Lleida
  - Hospital 12 de Octobre, Madrid
  - HCU Virgen de la Victoria, Málaga
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital Mutua de Terrassa, Terrassa (Barcelona)
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (3):
  - Lanssjukhuset Ryhov, Jönköping
  - Norrlands Universitetssjukhus, Umeå
  - Centrallasarettet Vasteras, Västerås
- United Kingdom (10):
  - Clatterbridge Centre for Oncology NHS Trust, Bebington, Wirral
  - Addenbrookes Hospital, Cambridge
  - Royal Surrey County Hospital, Guildford
  - Guy's and St Thomas' Hospital - London, London
  - St George's Hospital, London
  - Royal Marsden Hospital, London
  - Christie NHS Trust Hospital, Manchester
  - Nottingham City Hospital, Nottingham
  - Northern Lincolnshire and Goole Hospitals NHS Foundation Trust, Scunthorpe
  - Royal Marsden Hospital, Sutton

REFERENCES:
- [Background] Vogelzang NJ, Fizazi K, Burke JM, De Wit R, Bellmunt J, Hutson TE, Crane E, Berry WR, Doner K, Hainsworth JD, Wiechno PJ, Liu K, Waldman MF, Gandhi A, Barton D, Jungnelius U, Fandi A, Sternberg CN, Petrylak DP. Circulating Tumor Cells in a Phase 3 Study of Docetaxel and Prednisone with or without Lenalidomide in Metastatic Castration-resistant Prostate Cancer. Eur Urol. 2017 Feb;71(2):168-171. doi: 10.1016/j.eururo.2016.07.051. Epub 2016 Aug 10. PMID 27522164
- [Result] Petrylak DP, Vogelzang NJ, Budnik N, Wiechno PJ, Sternberg CN, Doner K, Bellmunt J, Burke JM, de Olza MO, Choudhury A, Gschwend JE, Kopyltsov E, Flechon A, Van As N, Houede N, Barton D, Fandi A, Jungnelius U, Li S, de Wit R, Fizazi K. Docetaxel and prednisone with or without lenalidomide in chemotherapy-naive patients with metastatic castration-resistant prostate cancer (MAINSAIL): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet Oncol. 2015 Apr;16(4):417-25. doi: 10.1016/S1470-2045(15)70025-2. Epub 2015 Mar 3. PMID 25743937
- [Result] de Morree ES, Vogelzang NJ, Petrylak DP, Budnik N, Wiechno PJ, Sternberg CN, Doner K, Bellmunt J, Burke JM, Ochoa de Olza M, Choudhury A, Gschwend JE, Kopyltsov E, Flechon A, van As N, Houede N, Barton D, Fandi A, Jungnelius U, Li S, Li JS, de Wit R. Association of Survival Benefit With Docetaxel in Prostate Cancer and Total Number of Cycles Administered: A Post Hoc Analysis of the Mainsail Study. JAMA Oncol. 2017 Jan 1;3(1):68-75. doi: 10.1001/jamaoncol.2016.3000. PMID 27560549

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following a safety and efficacy data review by the Data Monitoring Committee( DMC), the trial was stopped for futility. At that time, 1059 participants had been randomized and 1046 treated with either lenalidomide plus docetaxel and prednisone or placebo plus docetaxel and prednisone. A data cutoff date of 13 January 2012 was established.
Pre-assignment Details: Participants who had started a treatment cycle at the time of termination request were allowed to complete the cycle and have their discontinuation visit at the next cycle (21 days later). The safety follow-up of 28 days was also added to ensure all adverse events were followed.
Groups:
- Docetaxel/Prednisone/Placebo (DP): Participants received docetaxel 75 mg/m^2 by intravenous (IV) administration over 60 minutes on Day 1, prednisone 5 mg orally twice a day (BID) and identically matching placebo capsules daily (QD) on Days 1-14 in each 21-day treatment cycle.
- Docetaxel/Prednisone/Lenalidomide (DPL): Participants received docetaxel 75 mg/m^2 by intravenous (IV) administration over 60 minutes on Day 1, prednisone 5 mg orally twice a day (BID) and lenalidomide 25 mg capsules daily (QD) on Days 1-14 in each 21-day treatment cycle.
Period: Overall Study
Arm/Group | Docetaxel/Prednisone/Placebo (DP) | Docetaxel/Prednisone/Lenalidomide (DPL)
Started | 526 | 533
Treated | 521 | 525
Completed | 95 (DP Completed = kept on treatment with docetaxel/prednisone; Placebo was discontinued in DP arm) | 95 (DPL Completed = kept on treatment with docetaxel/prednisone; Lenalidomide discontinued in DPL arm)
Not Completed | 431 | 438
Not completed — Adverse Event | 71 | 122
Not completed — Disease Progression | 103 | 89
Not completed — Withdrawal by Subject | 50 | 57
Not completed — Death | 9 | 15
Not completed — Lost to Follow-up | 2 | 3
Not completed — Protocol Violation | 9 | 2
Not completed — Sponsor Decision | 102 | 78
Not completed — Clinical Progression | 17 | 16
Not completed — Biochemical Progression | 21 | 7
Not completed — Clinical Deterioration | 7 | 14
Not completed — Subject Decision/Investigator Discretion | 32 | 32
Not completed — Other | 8 | 3

BASELINE CHARACTERISTICS:
Population: Includes those from the Intent to Treat population (ITT). The ITT population is defined as all participants who were randomized, independent of whether they received study treatment or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel/Prednisone/Placebo (DP) | Docetaxel/Prednisone/Lenalidomide (DPL) | Total
Number analyzed (Participants) | 526 | 533 | 1059
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (7.79) | 68.9 (7.98) | 68.7 (7.89)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 171 | 163 | 334
  > = to 65 years and < = 75years | 246 | 244 | 490
  >75 years | 109 | 126 | 235
Sex/Gender, Customized [Number; unit: Participants]
  male | 526 | 533 | 1059
  female | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Rest of World includes Israel, Russia, Mexico and South Africa
  Participants
    US or Canada | 136 | 140 | 276
    EU or Australia | 329 | 330 | 659
    Rest of World (Includes 4 additional countries) | 61 | 63 | 124
Race, Customized [Count of Participants; unit: Participants]
  White | 433 | 436 | 869
  Other or no answer | 55 | 67 | 122
  Black or African American | 25 | 21 | 46
  Asian | 8 | 6 | 14
  American Indian or Alaska Native | 5 | 3 | 8
Weight [Mean (Standard Deviation); unit: kilograms] | 86.4 (16.18) | 86 (15.70) | 86.2 (15.93)
Height [Mean (Standard Deviation); unit: centimeters] | 174.0 (7.81) | 174.4 (7.38) | 174.2 (7.60)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — BMI or body mass index is a statistical benchmark that compares an individual's height and weight.
  kg/m^2 | 28.6 (5.02) | 28.3 (4.60) | 28.4 (4.81)
Body Mass Index, Categorical [Count of Participants; unit: Participants]
  <25 kg/m^2 | 134 | 138 | 272
  25-30 kg/m^2 | 221 | 243 | 464
  >30 kg/m^2 | 171 | 152 | 323
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a patient's disease is progressing, assess how the disease affects the daily living activities of the patient and determine appropriate treatment and prognosis.
  Participants
    0 (Fully Active) | 257 | 252 | 509
    1 (Restrictive but ambulatory) | 247 | 256 | 503
    2 (Ambulatory but unable to work) | 21 | 24 | 45
    3 (Limited self-care) | 1 | 0 | 1
    Not specified | 0 | 1 | 1
Type of Disease Progression [Count of Participants; unit: Participants] — Categories of specific indicators of disease progression type
  Participants
    Rising PSA only | 146 | 159 | 305
    Radiographic progression | 380 | 374 | 754
Prior Radiotherapy [Count of Participants; unit: Participants] — Participants who had been treated with prior radiation therapy
  Participants
    Yes | 308 | 312 | 620
    No | 218 | 221 | 439
Prior Cancer Surgery [Count of Participants; unit: Participants] — Participants who had undergone a surgical procedure associated with their prostate cancer diagnosis prior to study participation
  Participants
    Yes | 335 | 358 | 693
    No | 191 | 175 | 366
Other Prior Anti-Cancer Therapy [Count of Participants; unit: Participants] — Participants who were treated with other types of anti-cancer therapies prior to participation in study
  Participants
    Yes | 79 | 71 | 150
    No | 447 | 462 | 909
Baseline PSA (Prostate Specific Antigen) Levels [Mean (Standard Deviation); unit: (ng/ml)] — Prostate-specific antigen (PSA) is a substance produced by the prostate gland. Elevated PSA levels may indicate prostate cancer or a noncancerous condition such as prostatitis or an enlarged prostate.
  (ng/ml) | 290.359 (659.1583) | 316.501 (776.1133) | 303.542 (720.2895)
Metastatic Sites of Disease Outside of Prostate [Count of Participants; unit: Participants] — Specific sites of the body that have advanced spread of the prostate cancer.
  Participants
    Bone only | 157 | 169 | 326
    Soft tissues only | 94 | 104 | 198
    Both bone and Soft tissues | 273 | 259 | 532
    None | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was the time from the date of randomization to the date of death from any cause. If no death was reported for a participant before the cut-off date for OS analysis, OS was censored at the last date at which the participant was alive. The median OS was calculated based on Kaplan-Meier estimates and corresponding 95% confidence interval (CI) was calculated using the method provided by Brookmeyer and Crowley.
Time Frame: From randomization until death from any cause up to the cut-off date of 13 January 2012; up to approximately 26 months
Population: Intent-to-Treat (ITT) population defined as all randomized patients irrespective of whether they received treatment or not.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Docetaxel/Prednisone/Placebo (DP) | Docetaxel/Prednisone/Lenalidomide (DPL)
Number analyzed (Participants) | 526 | 533
weeks | NA [75.71 to NA] — Median overall survival was not reached for the DP arm as only 92 (17.5 %) of participants had died at the time of the data cut off. | 77 [64.29 to 81.71]
Statistical Analysis 1: Comparison: Docetaxel/Prednisone/Placebo (DP) vs Docetaxel/Prednisone/Lenalidomide (DPL); Test type: Superiority or Other; p = 0.0017, Log Rank — p-value is based on unstratified log-rank test; Hazard Ratio (HR) = 1.53, 95% CI 2-sided [1.17 to 2.00]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was the time from randomization to disease progression, or death, whatever occurred first. Progression criteria was met by analysis of target and non-target lesions as defined by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria. Progressive Disease (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters while on study or the appearance of one or more new lesions; an increase of at least 5mm as a total sum. Lymph nodes identified as target lesions (≥ 15 mm diameter in short axis) will be followed and reported by changes in diameter of short axis; or the unequivocal progression of a non-target lesion defined as an increase in the overall disease burden based on the change in non-measurable disease that is comparable in scope to the increase required to declare PD for measurable disease; Two or more new bone lesions as detected by bone scan
Time Frame: From randomization until disease progression or death from any cause; up to the cut-off date of 13 Jan 2012; maximum time on study was approximately 26 months
Population: Based on the Intent to treat population (ITT), defined as all randomized patients irrespective of whether they received treatment or not.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Docetaxel/Prednisone/Placebo (DP) | Docetaxel/Prednisone/Lenalidomide (DPL)
Number analyzed (Participants) | 526 | 533
Weeks | 46 [42.14 to 53.57] | 45 [38.0 to 46.14]
Statistical Analysis 1: Comparison: Docetaxel/Prednisone/Placebo (DP) vs Docetaxel/Prednisone/Lenalidomide (DPL); Test type: Superiority or Other; p = 0.0187, Log Rank; P-value is based on unstratified log-rank test; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [1.05 to 1.66]

3. Secondary Outcome: Percentage of Participants With an Objective Response According to Response Evaluation Criteria in Solid Tumors - RECIST Version 1.1 Criteria
Description: Objective response (OR) is defined as having complete response (CR) or partial response (PR) as best overall response based on RECIST Criteria 1.1 and defines a CR = Disappearance of all target lesions except lymph nodes (LN); LN must have a decrease in the short axis to <10mm; PR = 30% decrease in sum of diameters of target lesions taking as reference the baseline sum diameters; Progressed Disease (PD) = 20% increase in sum of diameters of target lesions taking as a reference the smallest sum of diameters and an absolute increase of ≥5 mm; the appearance of ≥1 new lesions; Stable Disease (SD)= Neither shrinkage to qualify for PR nor increase to qualify for PD taking the smallest sum diameters on study as reference. For non-target lesions a CR = Disappearance of all non-target lesions and all LN must be non-pathological in size <10 mm; Non-CR/Non PD: persistence of one or more non-target lesions; PD = unequivocal progression of existing non-target lesions or appearance of new ones
Time Frame: From day 1 to data cut-off 13 January 2012; maximum time on study was approximately 26 months
Population: Based on the ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel/Prednisone/Placebo (DP) | Docetaxel/Prednisone/Lenalidomide (DPL)
Number analyzed (Participants) | 526 | 533
percentage of participants | 24.3 | 22.1
Statistical Analysis 1: Comparison: Docetaxel/Prednisone/Placebo (DP) vs Docetaxel/Prednisone/Lenalidomide (DPL); Test type: Superiority or Other; p = 0.3975, Chi-squared; Odds Ratio (OR) = 0.884, 95% CI 2-sided [0.665 to 1.176]

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: A TEAE is defined as any AE occurring or worsening on or after the first dose of study drug and within 28 days after the last dose of study drug. A TESAE is defined as any serious adverse event (SAE) occurring or worsening on or after the first dose of study drug and within 28 days after the last dose of study drug. Safety and severity was assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0; Severity of AEs were graded (including second primary malignancies) as Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe; Grade 4- Life-threatening; Grade 5-Fatal;
Time Frame: From the time from of first dose of study drug administration to 28 days after the last dose of study drug and up to the data cut off date of 13 January 2012; the maximum duration of study drug was 93 weeks for DP and 90.6 weeks for DPL
Population: The Safety Population is defined as all randomized participants who receive at least one dose of the study treatment (lenalidomide/placebo, Docetaxel, or Prednisone).
Measure: Number; unit: participants
Arm/Group | Docetaxel/Prednisone/Placebo (DP) | Docetaxel/Prednisone/Lenalidomide (DPL)
Number analyzed (Participants) | 521 | 525
participants
  Any TEAE | 512 | 517
  Any TEAE related to lenalidomide or placebo | 379 | 412
  Any TEAE related to docetaxel/prednisone | 475 | 481
  Any severity grade 3-4 TEAE | 303 | 381
  Any serious AE (SAE) | 171 | 279
  Any SAE related to lenalidomide or placebo | 62 | 167
  Any SAE related to docetaxel/prednisone | 86 | 182
  Any AE causing discontinuation of lenalidomide/PBO | 82 | 150
  Any AE causing withdrawal of docetaxel/prednisone | 127 | 169
  Any TEAE leading to death | 16 | 24

5. Secondary Outcome: Percentage of Participants Who Received Post-Study Therapies
Description: Percentage of Participants Who Received Post-Study Therapies for advanced Prostate Cancer.
Time Frame: The date when the first consent form was signed to the last date of AE data collection;up to 5 years; up to the date of the final data analysis date of 20 April 2017
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Units Other Than Participants: Participants
Arm/Group | Docetaxel/Prednisone/Placebo (DP) | Docetaxel/Prednisone/Lenalidomide (DPL)
Number analyzed (Participants) | 521 | 525
Percentage of Participants | 70.8 | 69.0

6. Secondary Outcome: Percentage of Participants With Secondary Primary Malignancies During the Course of the Trial
Description: Second primary malignancies were monitored as events of interest and reported as serious adverse events throughout the course of the trial.
Time Frame: The date when the first consent form was signed to the last date of AE data collection; up to the date of the final data analysis date of 30 November 2016; 7 years and 19 days
Population: The Safety Population is defined as all randomized participants who receive at least one dose of the study treatment lenalidomide/placebo, Docetaxel, or Prednisone).
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel/Prednisone/Placebo (DP) | Docetaxel/Prednisone/Lenalidomide (DPL)
Number analyzed (Participants) | 521 | 525
percentage of participants
  Invasive Secondary Primary Malignancies | 1.3 | 1.7
  Non-invasive Secondary Primary Malignancies | 0.4 | 1.0

7. Secondary Outcome: Time to Onset of Secondary Primary Malignancies
Description: Time of Onset of Secondary Primary Malignancies was considered an event of interest
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Median (Full Range); unit: months
Arm/Group | Docetaxel/Prednisone/Placebo (DP) | Docetaxel/Prednisone/Lenalidomide (DPL)
Number analyzed (Participants) | 521 | 525
months | 29.7 [0.6 to 48.7] | 19.7 [3.7 to 65.0]

ADVERSE EVENTS:
Time Frame: From first dose of study treatment to 28 days after the last dose; as of the final analysis cut-off of 20 April 2017; median overall duration of treatment was 22.1 months for DPL and 27.0 months for the DP group
Groups:
- Docetaxel/ Prednisone/and Placebo (DP): Participants received Docetaxel 75 mg/m^2 by intravenous (IV) administration over 30-60 minutes on Day 1, Prednisone 5 mg orally twice a day (BID) and identically matching placebo capsules daily (QD) on Days 1-14 in each 21-day treatment cycle.
Arm/Group | Docetaxel/Prednisone/Lenalidomide (DPL) | Docetaxel/ Prednisone/and Placebo (DP)
Serious Adverse Events (participants affected / at risk) | 283/525 | 176/521
Other Adverse Events (participants affected / at risk) | 513/525 | 511/521
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel/Prednisone/Lenalidomide (DPL) (N=525) | Docetaxel/ Prednisone/and Placebo (DP) (N=521)
ANAEMIA (Blood and lymphatic system disorders) | 18 | 12
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 | 1
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 2 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 52 | 23
LEUKOPENIA (Blood and lymphatic system disorders) | 5 | 6
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 32 | 11
PANCYTOPENIA (Blood and lymphatic system disorders) | 4 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 2 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 2
ANGINA PECTORIS (Cardiac disorders) | 1 | 1
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0
ARRHYTHMIA (Cardiac disorders) | 2 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 14 | 8
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0
ATRIAL TACHYCARDIA (Cardiac disorders) | 1 | 1
ATRIAL THROMBOSIS (Cardiac disorders) | 1 | 0
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 0
BRADYCARDIA (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 2
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 0
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 0
CARDIOVASCULAR DISORDER (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 | 1
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 0 | 1
DILATATION VENTRICULAR (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 3 | 1
PALPITATIONS (Cardiac disorders) | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1
TACHYARRHYTHMIA (Cardiac disorders) | 1 | 0
TACHYCARDIA PAROXYSMAL (Cardiac disorders) | 0 | 1
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 1
MENIERE'S DISEASE (Ear and labyrinth disorders) | 1 | 0
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 1
ANAL FISTULA (Gastrointestinal disorders) | 0 | 1
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
ANAL ULCER (Gastrointestinal disorders) | 0 | 1
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 4 | 2
DIARRHOEA (Gastrointestinal disorders) | 22 | 5
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0
DIVERTICULUM (Gastrointestinal disorders) | 0 | 1
DUODENAL ULCER (Gastrointestinal disorders) | 1 | 0
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
ENTEROCOLITIS (Gastrointestinal disorders) | 1 | 0
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 1 | 0
FAECALOMA (Gastrointestinal disorders) | 1 | 0
FEMORAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 1 | 0
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 1 | 0
INTESTINAL INFARCTION (Gastrointestinal disorders) | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 | 2
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
MELAENA (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 4 | 2
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 0 | 2
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 4
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 1
SUBILEUS (Gastrointestinal disorders) | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2
VOMITING (Gastrointestinal disorders) | 8 | 3
ASTHENIA (General disorders) | 5 | 2
CHILLS (General disorders) | 1 | 0
DEATH (General disorders) | 0 | 1
DEVICE OCCLUSION (General disorders) | 0 | 2
FATIGUE (General disorders) | 4 | 2
GAIT DISTURBANCE (General disorders) | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 11 | 5
GENERALISED OEDEMA (General disorders) | 1 | 0
MALAISE (General disorders) | 1 | 0
MULTI-ORGAN FAILURE (General disorders) | 1 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 4 | 2
OEDEMA PERIPHERAL (General disorders) | 0 | 2
PAIN (General disorders) | 1 | 0
PERFORMANCE STATUS DECREASED (General disorders) | 1 | 0
PYREXIA (General disorders) | 19 | 6
THROMBOSIS IN DEVICE (General disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0
GALLBLADDER PERFORATION (Hepatobiliary disorders) | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 3 | 1
ABDOMINAL ABSCESS (Infections and infestations) | 0 | 1
ABSCESS BACTERIAL (Infections and infestations) | 1 | 1
ABSCESS JAW (Infections and infestations) | 1 | 0
ANAL ABSCESS (Infections and infestations) | 1 | 0
APPENDICITIS (Infections and infestations) | 1 | 0
APPENDICITIS PERFORATED (Infections and infestations) | 0 | 1
BACTERAEMIA (Infections and infestations) | 2 | 1
BRONCHITIS (Infections and infestations) | 2 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 0
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 1 | 1
CANDIDIASIS (Infections and infestations) | 1 | 0
CELLULITIS (Infections and infestations) | 3 | 3
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 2 | 0
DIARRHOEA INFECTIOUS (Infections and infestations) | 0 | 1
DIVERTICULITIS (Infections and infestations) | 1 | 0
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 | 0
ERYSIPELAS (Infections and infestations) | 0 | 1
ESCHERICHIA SEPSIS (Infections and infestations) | 1 | 1
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 1
GROIN ABSCESS (Infections and infestations) | 1 | 0
H1N1 INFLUENZA (Infections and infestations) | 1 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 0
HORDEOLUM (Infections and infestations) | 0 | 1
INCISION SITE CELLULITIS (Infections and infestations) | 0 | 1
INFECTIOUS PERITONITIS (Infections and infestations) | 1 | 0
INFECTIVE TENOSYNOVITIS (Infections and infestations) | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1
LUNG INFECTION (Infections and infestations) | 4 | 0
LYMPHANGITIS (Infections and infestations) | 0 | 1
NECROTISING FASCIITIS (Infections and infestations) | 1 | 0
NEUTROPENIC INFECTION (Infections and infestations) | 2 | 1
NEUTROPENIC SEPSIS (Infections and infestations) | 15 | 6
ORAL CANDIDIASIS (Infections and infestations) | 1 | 0
ORAL INFECTION (Infections and infestations) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 1 | 0
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 2 | 0
PNEUMONIA (Infections and infestations) | 24 | 8
PNEUMONIA BACTERIAL (Infections and infestations) | 0 | 1
PNEUMONIA INFLUENZAL (Infections and infestations) | 1 | 0
PNEUMONIA LEGIONELLA (Infections and infestations) | 1 | 0
PSEUDOMONAL BACTERAEMIA (Infections and infestations) | 1 | 1
PSEUDOMONAL SEPSIS (Infections and infestations) | 1 | 0
PYELONEPHRITIS (Infections and infestations) | 1 | 1
RECTAL ABSCESS (Infections and infestations) | 1 | 0
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1
RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 | 1
SEPSIS (Infections and infestations) | 3 | 9
SEPTIC SHOCK (Infections and infestations) | 3 | 1
SINUSITIS (Infections and infestations) | 1 | 0
SKIN INFECTION (Infections and infestations) | 2 | 0
STREPTOCOCCAL INFECTION (Infections and infestations) | 0 | 1
TONSILLITIS (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0
URETHRITIS (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 10 | 7
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 | 1
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION FUNGAL (Infections and infestations) | 0 | 1
UROSEPSIS (Infections and infestations) | 2 | 1
VESTIBULAR NEURONITIS (Infections and infestations) | 0 | 1
VIRAL INFECTION (Infections and infestations) | 1 | 0
WOUND INFECTION (Infections and infestations) | 0 | 1
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
TRAUMATIC LIVER INJURY (Injury, poisoning and procedural complications) | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 1 | 0
BLOOD UREA INCREASED (Investigations) | 1 | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 2 | 0
PLATELET COUNT DECREASED (Investigations) | 0 | 1
TROPONIN INCREASED (Investigations) | 1 | 0
URINE OUTPUT DECREASED (Investigations) | 0 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 13 | 4
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 | 1
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 | 1
GOUT (Metabolism and nutrition disorders) | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 2
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 3 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 | 0
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 2
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 4
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
FISTULA (Musculoskeletal and connective tissue disorders) | 1 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 2
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 1 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 1
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 2 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LYMPHOCYTIC LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTATIC PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SUPERFICIAL SPREADING MELANOMA STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 2 | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 3
DIZZINESS (Nervous system disorders) | 2 | 0
DYSKINESIA (Nervous system disorders) | 0 | 1
HYPOAESTHESIA (Nervous system disorders) | 1 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 2 | 0
LACUNAR INFARCTION (Nervous system disorders) | 1 | 0
PARKINSON'S DISEASE (Nervous system disorders) | 1 | 0
PRESYNCOPE (Nervous system disorders) | 1 | 0
SCIATICA (Nervous system disorders) | 1 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 | 3
SYNCOPE (Nervous system disorders) | 8 | 4
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 5 | 0
TREMOR (Nervous system disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 0 | 2
COMPLETED SUICIDE (Psychiatric disorders) | 1 | 0
DELIRIUM (Psychiatric disorders) | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 2
CALCULUS URETHRAL (Renal and urinary disorders) | 0 | 1
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 0 | 1
DYSURIA (Renal and urinary disorders) | 1 | 1
HAEMATURIA (Renal and urinary disorders) | 5 | 9
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 4
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 2
RENAL FAILURE (Renal and urinary disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 10 | 4
RENAL INJURY (Renal and urinary disorders) | 2 | 0
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 | 1
URETHRAL OBSTRUCTION (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 3 | 3
PELVIC PAIN (Reproductive system and breast disorders) | 0 | 1
PENILE HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ALVEOLITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 13 | 2
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 3 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 3 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 34 | 8
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DERMATITIS EXFOLIATIVE (Skin and subcutaneous tissue disorders) | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 | 1
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 13 | 3
EMBOLISM (Vascular disorders) | 1 | 1
HAEMATOMA (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 8 | 7
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 0 | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 | 2
THROMBOPHLEBITIS (Vascular disorders) | 2 | 0
VENA CAVA THROMBOSIS (Vascular disorders) | 1 | 0
VENOUS THROMBOSIS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel/Prednisone/Lenalidomide (DPL) (N=525) | Docetaxel/ Prednisone/and Placebo (DP) (N=521)
ANAEMIA (Blood and lymphatic system disorders) | 154 | 94
LEUKOPENIA (Blood and lymphatic system disorders) | 40 | 34
NEUTROPENIA (Blood and lymphatic system disorders) | 125 | 94
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 39 | 18
LACRIMATION INCREASED (Eye disorders) | 53 | 63
ABDOMINAL PAIN (Gastrointestinal disorders) | 55 | 36
CONSTIPATION (Gastrointestinal disorders) | 144 | 124
DIARRHOEA (Gastrointestinal disorders) | 236 | 204
DYSPEPSIA (Gastrointestinal disorders) | 41 | 30
NAUSEA (Gastrointestinal disorders) | 170 | 153
STOMATITIS (Gastrointestinal disorders) | 50 | 37
VOMITING (Gastrointestinal disorders) | 93 | 63
ASTHENIA (General disorders) | 124 | 117
FATIGUE (General disorders) | 238 | 232
MUCOSAL INFLAMMATION (General disorders) | 37 | 43
OEDEMA PERIPHERAL (General disorders) | 146 | 134
PYREXIA (General disorders) | 92 | 74
NASOPHARYNGITIS (Infections and infestations) | 46 | 37
URINARY TRACT INFECTION (Infections and infestations) | 36 | 32
WEIGHT DECREASED (Investigations) | 96 | 54
DECREASED APPETITE (Metabolism and nutrition disorders) | 125 | 105
DEHYDRATION (Metabolism and nutrition disorders) | 38 | 23
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 35 | 36
HYPOKALAEMIA (Metabolism and nutrition disorders) | 63 | 22
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 86 | 73
BACK PAIN (Musculoskeletal and connective tissue disorders) | 88 | 91
BONE PAIN (Musculoskeletal and connective tissue disorders) | 59 | 66
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 85 | 46
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 25 | 30
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 31 | 27
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 39 | 29
MYALGIA (Musculoskeletal and connective tissue disorders) | 44 | 55
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 57 | 66
DIZZINESS (Nervous system disorders) | 61 | 48
DYSGEUSIA (Nervous system disorders) | 113 | 124
HEADACHE (Nervous system disorders) | 42 | 51
PARAESTHESIA (Nervous system disorders) | 34 | 65
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 99 | 130
INSOMNIA (Psychiatric disorders) | 60 | 64
COUGH (Respiratory, thoracic and mediastinal disorders) | 108 | 76
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 104 | 88
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 37 | 52
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 30 | 20
ALOPECIA (Skin and subcutaneous tissue disorders) | 223 | 226
DRY SKIN (Skin and subcutaneous tissue disorders) | 39 | 50
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 22 | 32
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 41 | 59
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 14 | 28
PRURITUS (Skin and subcutaneous tissue disorders) | 46 | 10
RASH (Skin and subcutaneous tissue disorders) | 61 | 59
HYPERTENSION (Vascular disorders) | 16 | 33
HYPOTENSION (Vascular disorders) | 35 | 24

LIMITATIONS AND CAVEATS:
The independent DMC concluded that it was unlikely the trial would achieve its primary endpoint of improved overall survival. The sponsor agreed and the experimental lenalidomide/placebo treatment arm of the study was discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Multicenter publication must include input from investigators and Celgene, agreement to be established before publication. It has priority over subset (single center) publication, for duration of 24 months after study completion. Individual investigators have publication rights after multicenter publication is complete (or 24 months after study completion), whichever is first. In this case, Celgene has the right to comment and right to ask delay of publication for 60 days.